CLINICAL TRIAL: NCT02921646
Title: Monocentric, Prospective Study Assessing the Feasibility to Use Resting Energy Expenditure by Indirect Calorimetry as Prognostic Marker of Tumoral Response to 1st Line Chemotherapy in Patients Suffering From Metastatic Pancreatic Cancer
Brief Title: Relationship Between Evolution of Resting Energy Expenditure and Tumoral Response to Chemotherapy in Patients Suffering From Pancreas Cancer
Acronym: EnergiePancrea
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Protocol is not adapted to cancer pancreas disease as progression is very fast and patients stopped the study before 1st study assessment
Sponsor: Center Eugene Marquis (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2015-4-32-004
Record Dates: First submitted 2016-09-28; First posted 2016-10-03 (Estimated); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Metastatic Pancreatic Cancer
Keywords: energetic expenditure
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- energetic expenditure measure (Other): To a standard treatment by chemotherapy, energetic expenditure will be measured 5 times during the study.
  Interventions: Other: Measure of resting energetic expenditure

INTERVENTIONS:
Other: Measure of resting energetic expenditure — measure of resting energetic expenditure

SUMMARY:
The purpose of this study is to determine whether evolution of resting energetic expenditure is a predictive marker of tumoral response for patients suffering from metastatic pancreatic cancer and treated with 1st line of chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Pancreatic metastatic cancer
* Patient older than 18 years
* Initiation of a first line of chemotherapy by Folfirinox, or Gemcitabine or in combination with Nab-Paclitaxel.
* At least one measurable target lesion
* Patient signed consent for Energie-Pancreas study participation

Exclusion Criteria:

* Other concomitant cancer
* Major general status alteration ( Performance status = 3 or 4 at inclusion)
* Concomitant diseases explaining an altered general status or having an impact on energetic expenditure (i.e.chronic or severe infection, severe cardiac insufficiency, severe respiratory insufficiency, chronic inflammatory disease, recent surgery (< 1 month), ongoing Healing, hyperthyroidism.
* Smoker
* Patient deprived of his liberty, under guardianship, curator.
* Pregnant patient or breastfeeding
* Claustrophobic patient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-07-10 (Actual); Primary Completion 2019-07-10 (Actual); Study Completion 2019-07-10 (Actual)

PRIMARY OUTCOMES:
Resting energetic expenditure measurement by indirect calorimetry | 4 months
  Unit measure : calorie per day

CONTACTS AND LOCATIONS:
Overall Officials: Julien Edeline, MD, Principal Investigator — Centre Eugène Marquis
Locations (1):
- Centre Eugène Marquis, Rennes, France

IPD SHARING:
Plan to Share IPD: No